CLINICAL TRIAL: NCT03107000
Title: Corneal Endothelial Cell Loss After Trabeculectomy Versus Combined Trabeculectomy Phakoemulsification and IOL Implantation
Brief Title: Corneal Endothelial Cell Loss After Trabeculectomy Versus Phakotrabeculectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2915-001
Record Dates: First submitted 2017-01-18; First posted 2017-04-11 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Corneal Endothelial Cell Loss; Glaucoma
MeSH Terms: conditions — Corneal Endothelial Cell Loss; Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel group comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trabeculectomy group (Active Comparator): Patients with Open Angle Glaucoma requiring incisional surgery in whom specular microscopy can be performed without any delay in their treatment
  Interventions: Procedure: Trabeculectomy
- Phako-trabeculectomy group (Active Comparator): Patients with Open Angle Glaucoma and cataract requiring incisional surgery in whom specular microscopy can be performed without any delay in their treatment
  Interventions: Procedure: Phako-trabeculectomy

INTERVENTIONS:
Procedure: Trabeculectomy — Incisional surgery for glaucoma
  Other Names: Trab
  Arms: Trabeculectomy group
Procedure: Phako-trabeculectomy — Incisional surgery for glaucoma plus cataract
  Other Names: Phako-trab
  Arms: Phako-trabeculectomy group

SUMMARY:
Corneal endothelial cells health and pumping function is crucial to permit corneal optical clarity by keeping cornea in relatively dehydrated state. Corneal endothelial damage has been associated with most types of intraocular surgery. Trabeculectomy is the standard glaucoma surgical intervention in management of progressive glaucoma despite of medical therapy which can be performed in combination with Cataract surgery (Phacoemulsification and IOL implantation) in patients with cataract-impaired visual acuity.

In this study, the investigators will investigate and compare the corneal endothelial cells number and health status before and after trabeculectomy vs. combined surgery (at 1 month and 3 months post-op visits) using Specular microscopy which is a non-invasive technique to access the structure and function of the corneal endothelium by permitting visualization of the corneal endothelial mosaic to assess the effect of this surgical intervention on corneal endothelial cells health and number.

DETAILED DESCRIPTION:
Corneal endothelial cells health and pumping function is crucial to permit corneal optical clarity by keeping the cornea in a relatively dehydrated state.1 The corneal endothelium is a single layer of hexagonal cells with uniform size and shape in normal conditions. When endothelial cell density diminishes, the remaining cells increase in size to cover the empty spaces left by the dead cells, and therefore there is a change in the size (polymegathism) and morphology (pleomorphism) of the remaining cells. Trauma or other insults often cause endothelial cell death, which is irreparable because these cells lack division capacity.2,3,4 Corneal endothelial damage has been associated with most types of intraocular surgeries including glaucoma and cataract surgeries.5,6,7,8 Cataract and glaucoma are the most common causes of visual impairment worldwide.9,10

Phacoemulsification and Intraocular lens (IOL) insertion, the most commonly performed method of cataract extraction in the developed world, was first described in 1967.11 This technique allows rapid visual rehabilitation postoperatively and low induced astigmatism.11 The reported average loss of central corneal endothelial cells after phacoemulsification vary between 4% and 25%.8 Trabeculectomy, introduced by Cairns in 1968 12, is the most commonly performed incisional glaucoma procedure worldwide and has become the glaucoma filtering procedure of choice in glaucoma patients 5,13,14 with advanced glaucoma or poor tolerance or uncontrolled IOP despite of multiple topical or systemic medications with the goal of preserving vision and reducing the likelihood and rate of visual field loss and optic nerve changes in susceptible patients by reducing the intra ocular pressure (IOP) as the major risk factor.15,16 The use of anti-metabolites specifically Mitomycin C (MMC) as a supplement to trabeculectomy with more favorable effect on the outcome was reported by Chen 17 and Palmer 6 in the early 1990s5 showing eyes treated with MMC-augmented trabeculectomy have lower intraocular pressure (IOP) than eyes treated with trabeculectomy only.12 About 8.7% loss in central endothelial cells was reported after 3 months follow up in patients with Trabeculectomy with augmented Mitomycin C (MMC).7 Combined Trabeculectomy with Cataract surgery (Phacoemulsification and IOL insertion) can be performed based on the need to restore cataract-impaired visual acuity in trabeculectomy candidates.9,18 Given available results of previous studies on the effects of each of above mentioned procedures on corneal endothelial cells7,8, it is presumed that combined trabeculectomy with phacoemulsification and IOL insertion would have a cumulative effect on central corneal endothelial cell loss.

Specular microscopy is a non-invasive technique to assess the structure and function of the corneal endothelium by permitting visualization of the corneal endothelial mosaic.19 It is the standard method of endothelial cell analysis worldwide. By counting the number of the cells in measured areas of the cornea, an estimate of endothelial cell density can be made.

There is only one retrospective study available comparing central corneal endothelial cell loss after Trabeculectomy versus combined Trabeculectomy, Phacoemulsification and IOL insertion.2 There is also very limited data available to determine whether the expected damage is a non-progressive short-term effect or a progressive consequence which can lead to corneal endothelial decompensation. The investigator's aim is to evaluate and compare the effects of above mentioned procedures on central corneal endothelial cells health and density. The results of this study could help glaucoma surgeons make proper decisions in performing combined versus single surgeries in patients with initial risk factors for corneal decompensation.

3. Hypothesis The hypothesis of this study is that combined trabeculectomy, phacoemulsification and IOL implantation has more effect on corneal endothelial cell loss than trabeculectomy alone.

4. Research Plan 4.1 Study Design This is a prospective, interventional comparative clinical study

4.2 Patients Patients for this study will be recruited from the John and Liz Tory Eye Centre, Sunnybrook Health Sciences Centre (SHSC) in Toronto, Ontario, Canada. All patients will require and have consented to incisional glaucoma surgery with or without cataract surgery prior to being recruited. Subjects will be placed in one of two groups (Group A: Trabeculectomy only and Group B: Combined Surgery) based on absence or presence of cataract-impaired visual acuity. After achieving consent, for all patients undergoing the study, baseline information including age, gender, number of anti-glaucoma medications and medical history will be recorded. All patients will receive an ocular examination, including best corrected visual acuity measurement (Snellen chart), slit lamp examination along with tonometry (Goldmann applanation tonometry), central corneal thickness measurement (Pachymeter) and specular microscopy photos at pre-op, 1 month and 3 month visits. Anterior chamber depth will be measured by The IOLMaster® (Carl Zeiss Meditec, Jena, Germany) for all patients on pre-op visit. Type of the cataract will be assessed and recorded for Group B in pre-op visit. All achieved data will be recorded and saved on prepared data sheet for future analysis.

4.2-1 Inclusion criteria

1. Age over 18 years old
2. Patients with well established Open Angle Glaucoma (OAG) including Primary open angle glaucoma (POAG), Pseudoexfoliation Glaucoma (PXFG), Pigmentary Glaucoma (PG) and Steroid induced Glaucoma (SIG) requiring incisional surgery for IOP (Intraocular pressure) higher than target, despite receiving maximal tolerable medical treatment or were intolerant to medications with progressive glaucoma related visual field defects or optic nerve changes.
3. Patients with any of above types of glaucoma requiring cataract surgery.
4. Patients on which specular microscopy and IOLMaster can be performed without any delay in their treatment (availability of a qualified operator).
5. Decision makers able to give informed consent. 4.2-2 Exclusion criteria

1. Unable to attend follow -up visits 2. Angle closure glaucoma 3. Secondary open angle glaucoma other than PXFG, PG or SIG 4. Previous intraocular surgery or laser procedures other than laser trabeculoplasty 5. Post operative complications (if any) including flat anterior chamber, endophthalmitis and severe post op inflammation 6. Need to perform any other intraocular surgery during the course of the study 7. Pre-operation corneal disease

The investigators may decide to remove a patient from this study for any of the following reason(s):

• Need for any other ocular surgery known to have effects on corneal endothelial health

4.3 Surgical procedure

4.3 A: Trabeculectomy

The primary investigator and/or a glaucoma fellow will perform a standard trabeculectomy. After receiving a peribulbar block on identified eye, the patient will be transferred to OR and prepped and draped in the usual fashion.

A traction suture (6-0 silk) will be put in peripheral cornea after a lid speculum is inserted. A superior conjunctival peritomy will be performed followed by bipolar cautery for haemostasis. At this point 0.2 mg/ml Mitomycin-C will be applied using 3 soaked sponges tucked under conjunctival flap which will be removed after 90 seconds while checking the time by a digital timer. Copious irrigation with 20 cc sterile saline will be performed after.

A 4 in 4 mm scleral flap will be demarcated by a diamond blade at the depth of 0.25 mm. The flap will be elevated and dissected through the clear cornea using a crescent blade. After creating a side port to decompress the anterior chamber by a 25-gauge needle, sclerotomy will be performed using a 15 degrees blade followed by a peripheral iridotomy. The scleral flap will be sutured back into place using 4-8 interrupted and buried 10-0 nylon sutures.

Anterior chamber (AC) will be reformed by balanced sterile saline (BSS) which reveals filtration through the flap. Conjunctival flap will be repositioned meticulously into the limbus using either continuous alone or with combination of interrupted 8-0 Vicryl sutures. 6-0 silk traction suture and speculum will be removed after reforming AC again to confirm no leak from the wound site. The eye will be patched using an eye patch and a plastic shield after application of TobraDex® ointment and Atropine 1% eye drop (if Phakic).

4.3 B: Combined Trabeculectomy, Phacoemulsification and IOL implantation

The primary investigator and/or a glaucoma fellow will perform Combined trabeculectomy, phacoemulsification and IOL implantation. After receiving peribulbar block on identified eye, pt will be transferred to OR and prepped and draped in the usual fashion.

A traction suture (6-0 silk) will be put in peripheral cornea after a lid speculum is inserted. A superior conjunctival peritomy will be performed followed by bipolar cautery for haemostasis. At this point 0.2 mg/ml Mitomycin-C will be applied using 3 soaked sponges tucked under conjunctival flap which will be removed after 90 seconds while checking the time by a digital timer. Copious irrigation with 20 cc sterile saline will be performed after.

A 4 in 4 mm scleral flap will be demarcated by a diamond blade at the depth of 0.25 mm. The flap will be elevated and dissected through the clear cornea using a crescent blade.

After the side port is made using 15 degree blade, the entrance to the anterior chamber (AC) will be made using 2.4 mm keratome. Capsulorrhexis will be performed using a cyctotome after filling the anterior chamber with viscoelastic (Viscost® and Provisc®). Lens material will be extracted using phacoemulsification and completed by irrigation and aspiration of the cortex material. The capsular bag will be inflated using Provisc and Posterior Chamber Intra-Ocular Lens (PCIOL) will be inserted using the PCIOL dispenser in to the bag and dialed in place by a Sinskey hook. Completion of sclerotomy and creation of a peripheral iridectomy will be followed by using a 20 degree blade and Vannas scissors.

The scleral flap will be sutured back into place using 4-8 interrupted and buried 10-0 nylon sutures. AC will be reformed by balanced sterile saline (BSS) which reveals filtration through the flap. Conjunctival flap will be repositioned meticulously into the limbus using either continuous alone or with combination of interrupted 8-0 Vicryl sutures. 6-0 silk traction suture and speculum will be removed after reforming AC again to confirm no leak from the wound site. The eye will be patched using an eye patch and a plastic shield after application of TobraDex® ointment.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 y/o.
2. Patients with well established Open Angle Glaucoma including Primary open angle glaucoma, Pseudoexfoliation or Pigmentary Glaucoma & Steroid induced Glaucoma requiring incisional surgery for Intraocular pressure higher than target, despite receiving maximal tolerable medical treatment or were intolerant to medications with progressive glaucoma related visual field defects or optic nerve changes.
3. Any of a above who needs cataract surgery
4. In those specular microscopy can be performed without any delay in their treatment.
5. Decision makers able to give informed consent.

Exclusion Criteria:

1. Unable to attend follow -up visits.
2. Angle closure glaucoma.
3. Secondary open angle glaucoma other than PXFG, PG or SIG.
4. Previous intraocular surgery/laser procedures other than laser trabeculoplasty.
5. Post operative complications (if any) including flat anterior chamber, endophthalmitis & severe post op inflammation.
6. Pre-op corneal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Endothelial cell count | 3 months post surgery
  Specular microscopy

SECONDARY OUTCOMES:
IOP | 3 month visit
  Goldmann tonometry
Visual acuity | 3 month visit
  Snellen Acuity
Endothelial cell morphology - qualitative | 3 month visit
  Specular microscopy
Central corneal thickness | 3 month visit
  Ultrasound pachymetry

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Birt, MD, Principal Investigator — Sunnybrook Health Science Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No